CLINICAL TRIAL: NCT00700076
Title: Pilot Study of ORG 25935 Modulation of Ketamine-induced Behavioral and Cognitive Effects in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Organon (Industry)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Associate Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0701002174
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: ORG 25935; Ketamine; healthy subjects
MeSH Terms: interventions — Ketamine; N-methyl-N-(6-methoxy-1-phenyl-1,2,3,4-tetrahydronaphthalen-2-ylmethyl)aminomethylcarboxylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Ketamine and Org 25935
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo and Ketamine

INTERVENTIONS:
Drug: Ketamine and Org 25935 — Oral administration of Org 25935 16 mg and intravenous administration of ketamine (0.23 mg/kg bolus over 1 minute, followed by 0.58 mg/kg/hour x 30 minutes, followed by 0.29 mg/kg/hour x 69 minutes)
  Arms: 1
Drug: Placebo and Ketamine — Oral administration of placebo and intravenous administration of ketamine (0.23 mg/kg bolus over 1 minute, followed by 0.58 mg/kg/hour x 30 minutes, followed by 0.29 mg/kg/hour x 69 minutes)
  Arms: 2

SUMMARY:
Org 25935 is a new putative antipsychotic agent developed by N.V. Organon.The primary objective of this study is to investigate the effect of Org 25935 on ketamine-induced impairments in immediate recall.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18 - 55 years

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to the drugs used in the study or chemically related compounds or excipients which may be employed in the study or to any other unknown drug used in the past.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01-22 (Actual); Primary Completion 2009-03-09 (Actual); Study Completion 2009-03-09 (Actual)

PRIMARY OUTCOMES:
Attenuation of ketamine-induced cognitive deficits by Org 25935 | +20 to +100 minutes

SECONDARY OUTCOMES:
Attenuation of ketamine-induced schizophrenia-like psychotic symptoms, perceptual alterations, subjective high and deficits in attention and working memory by Org 25935. | 0 to +100 minutes
Investigation of interaction of polymorphisms of candidate genes e.g., BDNF, COMT with the effect of Org 25935 on ketamine induced psychotomimetic and amnestic deficits. | 0 to +100 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, M.D., Principal Investigator — Yale University School of Medicine, Department of Psychiatry
Locations (1):
- Biological Studies Unit at the VA Connecticut Healthcare System, Yale School of Medicine, West Haven, Connecticut, United States